CLINICAL TRIAL: NCT05282017
Title: LatInamerican Vaccine Effectiveness Against Hospitalizations Due to Circulating COVID-19 VoC RWE Study
Acronym: LIVE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8111R00016
Record Dates: First submitted 2022-02-18; First posted 2022-03-16 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-03

CONDITIONS: COVID-19, SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For those participating on the control group (previous positive PCR/antigen test) a new COVID-19 PCR test will be performed to evaluate the type of variant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: Meets the COVID-19 like case definition AND Tests positive for at least one SARS-CoV-2 RT-PCR test or Quick-Test (Antigen) with specimens collected between 14 days prior to and including within 24 hours of the day of hospital admission (day 0).
- Control Group: Meets the COVID-19 case definition AND Tests negative for all SARS-CoV-2 RT-PCR or Quick-Test (Antigen) tests with specimens collected between 14 days prior to and including a negative test the day at hospital admission (day 0).

SUMMARY:
COVID-19 is the infectious disease caused by the novel coronavirus known as SARS-CoV-2, that appeared in 2019. The World Health Organisation (WHO) declared the novel coronavirus a pandemic on 11 March 2020. The evolution of the pandemic is varying across countries, affected in part by different containment strategies ranging from extreme lockdown to relative inaction. As a result, there are regional waves of the disease and pockets of vulnerable populations. Globally, governments have acknowledged that effective vaccines against COVID-19 are the only way to guarantee a safe and sustained exit strategy from repeated lockdowns.

The objective of this study is to estimate the vaccine effectiveness against hospitalizations due to circulating COVID-19 VoC among subjects eligible for vaccination with the AstraZeneca or any other COVID-19 vaccine provided in their country as per national/regional immunization recommendations prior to hospital admission.

The study design is an observational prospective active-surveillance hospital-based study, with a test-negative case-control design (TNCC) of hospitalized COVID-19 like cases undergoing testing for SARS-CoV-2

DETAILED DESCRIPTION:
LatInamerican Vaccine Effectiveness against hospitalizations due to circulating COVID-19 VoC RWE study is an observational prospective active-surveillance hospital-based study, with a test-negative case-control design (TNCC) of hospitalized COVID-19 like cases undergoing testing for SARS-CoV-2 by RT-PCR or rapid antigen test with the participation of countries from six LatAm Marketing Companies (Argentina, Brazil, Colombia, Costa Rica, Mexico and Panama).

This study will generate new information regarding vaccine effectiveness (VE) in the RW setting for populations where evidence is still unavailable

ELIGIBILITY:
Inclusion Criteria:

* 18y and older
* Ever eligible for vaccination with the AstraZeneca or any other COVID-19 vaccine provided in their country as per national/regional immunization recommendations prior to hospital admission.
* Hospitalization due to COVID-19 like case
* Willing and able to provide informed consent (or by legal accepted representative if patient are not able to provide their signature by themselves)

Exclusion Criteria:

* Cannot be swabbed or other conditions that contra-indicate swabbing
* COVID-19 hospitalization within 3 months prior to the current admission. Hospital transfers are not considered as a prior hospitalization.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects older than 18y that are hospitalized due COVID-19 like symptoms
Sampling Method: Probability Sample
Enrollment: 792 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Number of hospitalized patients due COVID-19 like symptoms | From enrollment date until study completion, an average 1 year
  The outcome of interest for the primary analysis will be SARS-CoV-2 in patients hospitalized with/because of COVID-19 like symptoms

SECONDARY OUTCOMES:
SARS-CoV-2 variants detection | Through study completion and data analysis, an average of 1.5 year
  Include detection of SARS-CoV-2 genetic variants in test-positive cases.

OTHER OUTCOMES:
Disease severity (based on WHO severity scale, ICU admission, need of hemodialysis, mechanical ventilation) (Exploratory outcome) | From date of randomization until hospital discharge or date of death from any cause, whichever came first assessed up to 6 months
  Severity of hospitalization disease due to laboratory confirmed SARS-CoV-2 disease

CONTACTS AND LOCATIONS:
Locations (9):
- Brazil (3):
  - Research Site, Brazil, Rio de Janeiro
  - Research Site, Brazil, Salvador
  - Research Site, Brazil, São Paulo
- Colombia (2):
  - Research Site, Bogotá
  - Research Site, Cali
- Research Site, San José, Costa Rica
- Mexico (2):
  - Research Site, Guadalajara, Jalisco
  - Research Site, Mérida, Yucatán
- Research Site, Panama City, Panama

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles.
  For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Clinical Study Report (CSR) Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8111R00016&attachmentIdentifier=51f3eb0c-bbe2-405d-9065-99957b7e2287&fileName=Clinical_Study_Report_(CSR)_Synopsis.pdf&versionIdentifier=